CLINICAL TRIAL: NCT02140879
Title: LA Moms and Babies Study (LAMBS) for Nutrition and Growth
Acronym: LAMBS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB closed on 9/5/2018
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PBRC 11031
Record Dates: First submitted 2014-04-24; First posted 2014-05-16 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy; Inflammation
Keywords: pregnancy; inflammation; infant assessment
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsule 1 (Placebo Comparator): Placebo is a mixture of corn and soy oils.
  Interventions: Dietary Supplement: Capsule 1 or Capsule 2; Dietary Supplement: Capsule 2
- Capsule 2 (Active Comparator): Active supplement group, will take capsules containing oil '2' which is an algal oil.
  Interventions: Dietary Supplement: Capsule 1 or Capsule 2; Dietary Supplement: Capsule 2

INTERVENTIONS:
Dietary Supplement: Capsule 1 or Capsule 2 — Capsules will be consumed on a daily basis during pregnancy. One group, the placebo group of the study, will take capsules (2/day) containing oil '1 ' which is a mixture of corn and soy oils . The other group, the supplement group, will take capsules containing oil '2' which is an algal oil. Both oils are found in our diets.
Dietary Supplement: Capsule 2 — Two capsules will be consumed on a daily basis during pregnancy. The other group, the supplement group, will take capsules containing oil '2' which is an algal oil. Both oils are found in our diets. One group, the placebo group of the study, will take capsules containing oil '1 ' which is a mixture of corn and soy oils .

SUMMARY:
This research study will examine how diet during pregnancy can benefit pregnancy and pregnancy outcome, such as your baby's weight. More specifically, the investigators will study the effects of two different food oils/fats that are commonly consumed to determine if one is more effective in limiting maternal inflammation during pregnancy. You are being asked to take part in this study because it will help us update and make the best dietary recommendations for pregnant women and women of child bearing ages.

DETAILED DESCRIPTION:
Pregnant women will be asked to consume dietary supplements (2 capsules, from the Pennington Biomedical Pharmacy) each day during pregnancy. They will begin taking the capsules around 17 weeks of pregnancy and take them each day until their babies are born. Women will be randomized to one of two groups. Randomization means they will be put into a group by chance, similar to flipping a coin. One group, the placebo group of the study, will take capsules containing oil '1 ' which is a mixture of corn and soy oils . The other group, the supplement group, will take capsules containing oil '2' which is an algal oil. Both oils are found in our diets. Neither the subject nor the study staff will know which group women are in.

Women will also keep a diary of how many capsules they take. At around 17, 22, 24, 26, 30, 32, and 36 weeks of pregnancy, women will go to Woman's Hospital to get new capsules and return any remaining capsules and their capsule diary. If they are not able to go to Woman's Hospital at weeks 22, 26, or 32 a researcher will arrange to meet them at an agreed upon prearranged place, such as a pharmacy, a library, or Pennington Biomedical, for example. At the same visits to Woman's Hospital at weeks 17, 24, 30, and 36 weeks of pregnancy women will also have their blood drawn (approximately one tablespoon).

At 17, 22, 24, 26, 30, 32 and 36 weeks of pregnancy we will also ask women about the foods they are eating. We will do this by a prearranged phone call; women will not need to meet us in person for this.

Researchers will contact subjects weekly by phone to inquire about compliance with consumption of capsules. Contact will only take place during weeks in which a visit or phone call regarding diet is not required.

At 17, 24, 30, and 36 weeks of pregnancy small blood samples will be collected from their arm (approximately one tablespoon at each collection) for laboratory analyses. At the birth of their baby a sample of blood will be collected from the umbilical cord after their baby is delivered. All blood samples will be stored at Pennington Biomedical. Blood samples will be analyzed by the researchers who are involved in the study. Some analyses will take place at Pennington Biomedical and Louisiana State University (LSU). Deidentified (without subject names) samples will be sent to study researchers at Northeastern University in Boston, LSU Health Sciences Center in New Orleans, and DSM Nutritional Products in Columbia, Maryland for some of the analyses. At the end of the study remaining blood samples will be discarded unless women consent for their blood to be used for future research. Should women decide to withdraw from the study, any samples collected thus far will be included in the study since they will be deidentified and the investigators will not know which samples belong to each person. We will also collect information about the baby's birth weight, length, and health from the baby's hospital chart.

When the baby is 2 weeks, 6 months, and 12 months of age we will measure the baby's body fat and lean tissue. To do this measurement the baby will lie or sit in an enclosed chamber where the mother can see her baby during the measurements. There are no attachments made to the baby. At these times we will also determine the baby's body fat by measuring the thickness of the baby's skinfold; this is done by gently lifting a double fold of skin on the baby's hip, upper arm (triceps), and back of the thigh and measuring the thickness of that fold with a handheld instrument with two hinged arms that fit over the skinfold. There is no discomfort associated with this procedure. The measurements will be made at Woman's Hospital. During these visits we will also ask questions about how the mother is feeding her baby. Between these visits (when the baby is 2, 4, 8, and 10 months old) we will phone to ask about how the baby is being fed and to inquire about the mother's and baby's well-being.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy
* Caucasian/White and African-American ethnicities
* Between the ages of 18 and 35 years
* Overweight before becoming pregnant (BMI=25.0-29.9 kg/m2)
* Pass on the glucose tolerance test for diabetes

Exclusion Criteria:

* Have more than 5 children
* Have a history of high blood pressure, high blood lipids, kidney or liver disease
* Have inability to handle blood sugar normally
* Have polycystic ovary syndrome
* Have thyroid disorder
* Have multiple fetuses, pregnancy related complications (preterm labor; diagnosed with gestational diabetes mellitus, pregnancy impaired glucose tolerance, preeclampsia, a first degree relative with diabetes, gave birth to a previous large for gestational age infanthigh blood pressure, premature rupture of the membranes)
* Have smoked in the past 6 months
* Have been pregnant or lactating (breastfeeding) in the past year
* Do not want their baby's body fat measured throughout the first year of life
* Do not bring their prenatal record and study information copies to Woman's Hospital for delivery
* Deliver at a hospital other than Woman's Hospital
* Test positive for human immunodeficiency Virus (HIV), syphilis, sepsis, group B streptococcus, Hepatitis B
* Do not follow study procedures
* Planning to bank cord blood or unwilling to donate cord blood
* Planned/elective C-section.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Differences in maternal inflammation between the two study groups. | The Participant will be followed during pregnancy, between the 17th and 36th week of pregnancy, on average of 19 weeks.
  Pregnancy creates a state of insulin resistance that is worsened by excess weight during pregnancy and it is accompanied by inflammation. Inflammation in pregnant women will be measured by a blood draw from the arm and analysis of the blood.

SECONDARY OUTCOMES:
Differences in infant growth will be determined with measurements of infant height and weight and with an instrument that determines air displaced by the baby's body. | The participant will be followed the First year of life, an expected average of 52 weeks.
  Measurements of the baby will be calculated in an enclosed chamber where the baby will lie on a tray in a bassinet-like crib with a plastic cover where the baby will be able to see his mother. There will be no attachments to the baby. At these time periods the baby's body fat will also be measured by the thickness of the baby's skinfold; this is done by gently lifting a double fold of skin on the baby's hip, upper arm (triceps), and back of the thigh and measuring the thickness of that fold with a handheld instrument with two hinged arms that fit over the skinfold. There is no discomfort associated with this procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Lammi-Keefe, PhD, RD, Principal Investigator — PBRC
Locations (1):
- Womans Hospital, Baton Rouge, Louisiana, United States